CLINICAL TRIAL: NCT02516293
Title: Cardiac Rehabilitation Program in Patients With Chagas Heart Failure: a Pilot Study
Brief Title: Cardiac Rehabilitation in Chagas Heart Failure
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Evandro Chagas National Institute of Infectious Disease (Other)
Responsible Party: Principal Investigator, Mauro Felippe Felix Mediano, Clinical Researcher in Public Health, Evandro Chagas National Institute of Infectious Disease
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAAE 0055.0.009.000-11
Record Dates: First submitted 2015-07-31; First posted 2015-08-05 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Chagas Disease; Chagas Cardiomyopathy
MeSH Terms: conditions — Chagas Disease; Chagas Cardiomyopathy | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention group (Experimental): * Physical exercise intervention
  * Nutritional counseling
  * Pharmaceutical counseling
  Interventions: Behavioral: Exercise, nutritional and pharmaceutical counseling

INTERVENTIONS:
Behavioral: Exercise, nutritional and pharmaceutical counseling — Physical exercise intervention protocol was performed three times per week, 60 minutes per session, during 8 months. Exercise sessions consisted of 30 minutes of aerobic exercise on a treadmill or on a cycle ergometer, 20 minutes of strength exercises for the major muscle groups (sit-ups, push-ups, and pull-ups), and 10 minutes of stretching exercises. Nutritional and pharmaceutical consisted on general guidance about adequate eating habits for patients with heart failure, mainly sodium and water intake, and medication usage, particularly drug dosage and compliance.

SUMMARY:
Due to the lack of information in the literature about the role of cardiac rehabilitation on Chagas heart failure, the aim of the present study was to evaluate the effects of a cardiac exercise program on functional capacity, cardiac function, respiratory muscle strength, body composition, biomarkers and quality of life among Chagas heart failure patients.

DETAILED DESCRIPTION:
The present study consisted in a pre/post single-arm intervention study conducted at the Evandro Chagas National Institute of Infectious Disease (INI), located on Rio de Janeiro, Brazil. INI is a national reference center for treatment and research in infectious diseases and tropical medicine in Brazil, which follows a large cohort of patients with Chagas disease, all of them diagnosed by two simultaneously positive serological tests (enzyme-linked immunosorbent assay and indirect immunofluorescence). Patients included in the study were submitted to a physical exercise intervention protocol performed three times per week, 60 minutes per session, during an 8-month period. Nutritional and pharmaceutical counseling were also monthly provided during the follow-up and consisted on general guidance about adequate eating habits for patients with heart failure, mainly sodium and water intake, and medication usage, particularly drug dosage and compliance.Patients included in the study were followed during an 8-month period in which evaluations of functional capacity (maximal progressive cardiopulmonary exercise test), muscle respiratory strength (manovacuometry) and body composition (anthropometry and skinfolds) were performed at baseline, after four months and at the end of follow-up. Assessments of cardiac function (bidimensional echocardiography), biomarkers (lipid profile, glucose and glycated hemoglobin) and quality of life (Minnesota Living with Heart Failure questionnaire) were taken at baseline and after eight months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients at the stages C or D of Chagas cardiomyopathy
* Patients receiving standard optimized medical therapy
* Patients with good adherence to outpatient treatment within the last three months.

Exclusion Criteria:

* Those who were not able to attend three weekly training sessions,
* Those who had neuromuscular limitations, cardiopathies from non-Chagasic etiology (e.g ischemic), systemic conditions that limits exercise practice (e.g chronic obstructive pulmonary disease)
* Practitioners of regular exercise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-05; Primary Completion 2014-01 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Functional Capacity (VO2 max) | Change from baseline at 4 and 8 months
  VO2 max (ml/kg/min)

SECONDARY OUTCOMES:
Muscle respiratory strength (maximal inspiratory pressure and maximal expiratory pressure) | Change from baseline at 4 and 8 months
  Maximal inspiratory pressure and maximal expiratory pressure (cm H2O)
Body composition (body fat percentage) | Change from baseline at 4 and 8 months
  Body fat percentage (%)
Cardiac function (mainly ejection fraction) | Change from baseline at 8 months
  Ejection fraction (%)
Biomarkers (lipid profile and glucose) | Change from baseline at 8 months
  Total cholesterol, Triacylglycerol, HDL-cholesterol, LDL-cholesterol, VLDL-cholesterol (mg/dl) and glucose (mg/dl)
Biomarkers (glycated hemoglobin) | Change from baseline at 8 months
  Glycated hemoglobin (%)
Quality of life by Minnesota Living with heart failure questionnaire (MLHFQ) | Change from baseline at 8 months
  MLHFQ Score ranging from 0 to 105
Anthropometry | Change from baseline at 4 and 8 months
  Body weight (kg)
Anthropometry | Change from baseline at 4 and 8 months
  Waist and hip circumference (cm)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea S Sousa, PhD, Principal Investigator — Evandro Chagas National Institute of Infectious Disease
Locations (1):
- Evandro Chagas National Institute of Infectious Disease, Rio de Janeiro, Rio de Janeiro, Brazil